CLINICAL TRIAL: NCT04210609
Title: Treating Non-healing Foot Wounds With Vaporous Hyperoxia Therapy as an Adjunct to Standard Wound Care
Brief Title: Effectiveness of Vaporous Hyperoxia Therapy (VHT) in the Treatment of Chronic Diabetic Foot Ulcers
Acronym: VHTDFU2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vaporox (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAPOROX-VHT100-02
Record Dates: First submitted 2019-12-19; First posted 2019-12-24 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- VHT treatment (Experimental): Patients will be treated with VHT for 55 minutes at a minimum frequency of 2 times per week
  Interventions: Device: Vaporous Hyperoxia Therapy

INTERVENTIONS:
Device: Vaporous Hyperoxia Therapy — 55 minutes of treatment, 2 times per week
  Other Names: VHT

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Vaporous Hyperoxia Therapy (VHT) for the treatment of Diabetic Foot Ulcers.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effectiveness of Vaporous Hyperoxia Therapy (VHT) for the treatment of Diabetic Foot Ulcers. VHT treatments will be provided as an adjunct to standard wound care. Subjects will receive VHT treatments until wound closure, or for the treatment period of 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic foot wound, graded by the Wagner Scale as a 1,2 or 3
* Wound has resisted healing with standard wound care for at least 6 weeks
* No symptoms of sepsis
* Able to maintain reasonable nutrition and hydration
* Able to maintain adequate home care between treatment visits
* Able to understand and follow basic wound care instructions, or has caregiver who can assist

Exclusion Criteria:

* Skin wounds cancer/neoplastic etiology
* Wounds that involve osteomyelitis or tendon involvement
* Diagnosis of methicillin resistant staph aureus by wound swab
* Acute skin conditions
* Surgery within 30 days of study onset
* Wounds where the end cannot be probed
* Participation in another clinical trial within 120 days prior to study onset
* Non-compliant patients
* Pregnancy
* Presence of co-morbid conditions that in the physician's opinion exclude the individual from the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-10-03 (Estimated); Study Completion 2022-10-03 (Estimated)

PRIMARY OUTCOMES:
Wound closure rate at 20 weeks | 20 weeks
  The percentage of subjects that achieved complete wound closure by week 20, where wound closure is defined by complete re-epithelialization without drainage

SECONDARY OUTCOMES:
Wound closure rate at 12 weeks | 12 weeks
  The percentage of subjects that achieved complete wound closure by week 12, where wound closure is defined by complete re-epithelialization without drainage
Time to 50%, 75%, 100% wound closure | Up to 20 weeks
  Time to percent reduction in volume (length x width x depth) from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Dustin Kruse, DPM, Principal Investigator — Rocky Mountain Foot and Ankle Center
Locations (3):
- United States (3):
  - Rock Canyon Foot and Ankle Clinic, Castle Rock, Colorado
  - Rocky Mountain Foot and Ankle Center, Denver, Colorado
  - Colorado Foot and Ankle, Denver, Colorado